CLINICAL TRIAL: NCT06073912
Title: Simultaneous Implant Placement With Autogenous Corticocancellous Bone Block vs Mineralized Plasmatic Matrix in Maxillary Sinus Lifting (Randomized Clinical Trial)
Brief Title: Implant Placement With Corticocancellous Bone Block vs Mineralized Plasmatic Matrix in Maxillary Sinus Lifting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Abdel Salam Ibrahim Omara, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12323
Record Dates: First submitted 2023-08-14; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Maxillary Sinus Floor Elevation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autogenous corticocancellous block (Experimental): Autogenous bone graft harvested as a block from the chin area
  Interventions: Procedure: Open sinus lifting; Procedure: Collecting blood sample; Procedure: Bone graft harvesting; Procedure: Autogenous corticocancellous block graft; Device: Centrifuge
- Mineralized plasmatic matrix (Active Comparator): Mix of patient's PRP and autogenous particulate graft
  Interventions: Procedure: Open sinus lifting; Procedure: Collecting blood sample; Procedure: Bone graft harvesting; Procedure: Mineralized plasmatic matrix graft; Device: Centrifuge; Device: ACM bur

INTERVENTIONS:
Procedure: Open sinus lifting — Sinus lateral window to graft the floor of the sinus using sinus red diamond stone
Procedure: Collecting blood sample — Blood sample is collected to harvest PRP and PRF
Procedure: Bone graft harvesting — Bone graft harvesting from the chin area
Procedure: Autogenous corticocancellous block graft — Simultaneous implant placement with sinus lifting and grafting using autogenous corticocancellous block, stabilized inside the sinus using clamp or screws that will be removed before closure
  Arms: Autogenous corticocancellous block
Procedure: Mineralized plasmatic matrix graft — Simultaneous implant placement with sinus lifting and grafting using mineralized plasmatic matrix that is formed using PRP of the patient mixed with particulate autogenous graft from the chin area
  Arms: Mineralized plasmatic matrix
Device: Centrifuge — Centrifuge will be needed to get the PRP in the Comparator group and PRP in both groups
Device: ACM bur — Auto Chip Maker will be used to collect the autogenous particulate bone graft for the sticky bone graft
  Arms: Mineralized plasmatic matrix

SUMMARY:
Maxillary sinus floor elevation is a predictable and effective procedure for increasing the height of the residual bone in the posterior maxilla. The sinus lift procedure is basically performed using Conventional lateral sinus floor elevation (CLSFE) when RBH < 5 mm.

The use of autogenous corticocancellous bone block allows the simultaneous placement of an implant in the severely atrophic maxilla. Autogenous corticocancellous block will be applied in these patients to decrease the number of surgical interventions and the complications related to the surgery, without any additional risk, as well as to provide graft stabilization with the implant itself, using a mechanism similar to that of a screw and nut. Although the traditional application of sticky bone inside the sinus gives the benefit of moldable shaping and accurate fit into the recipient bony cavity which hardens and allows for implant osteotomy and installation with adequate implant stability. Limited comparative studies of both techniques had been introduced to the literature. This study is aimed to compare the quantity of bone gain after open sinus lift and augmentation using autogenous corticocancellous bone blocks from the chin area versus autogenous particulate mineralized plasmatic matrix (sticky bone) graft used as control group.

The primary outcome which is amount of bone gain will be measured and secondary stability of the implant.

DETAILED DESCRIPTION:
After meeting the inclusion criteria, A preoperative digital panoramic radiograph with 1:1 magnification will be taken for each patient as a primary survey in order to exclude the presence of any lesions at the area of interest. A cone beam computed tomography (CBCT) scan will be done to measure the amount of the remaining alverolar bone height preoperatively.

The procedure will start in both groups with administration of general anesthesia or local anesthesia PSA Nerve block, infraorbital block and greater palatine will be administered using mepivacaine HCl (2%) with levonordefrin 1:20 000 (Scandonest 2%; Septodont, Saint- Maur-des-Fossés, France) injection to control pain and bleeding. Scrubbing and draping of the patient will be carried out in a standard fashion using betadine.

Both groups will have open sinus lifting with simultaneous implant placement with different augmentation techniques.

The inte group will have autogenous corticocancellous block graft, while the comparator group will have mineralized plasmatic matrix (sticky bone) graft.

Autogenous bone graft will be harvested in both groups from the chin area, corticocancellous block (intervention group) and particulate chips (comparator group).

Blood sample will be collected from the patient in both groups. Bone graft will be stabilized in place during the drilling procedure using a clamp\screws.

Lateral window will be closed in both groups using PRF membrane.

ELIGIBILITY:
Inclusion Criteria:

* Patients with edentulous vertically deficient posterior maxillary ridge with remaining alveolar ridge bone height <4=/ mm.
* Both males as well as females without any active periodontal disease.
* All patients are in a good health with no systemic, immunologic, or debilitating diseases that could affect normal bone healing.
* Patients are free from T.M.J troubles, abnormal oral habits such as bruxism.
* The edentulous ridges are covered with optimal thickness of mucoperiosteum with no signs of inflammation, ulceration or scar tissue.
* Remaining natural teeth have good periodontal tissue support and occlusion showed sufficient inter arch space for future prosthesis.

Exclusion Criteria:

* On the local level, patients with maxillary sinus diseases, former sinus surgery and unfavorable inter maxillary relationship will be excluded.
* General contraindications to implant surgery.
* Remaining ridges>5mm
* Subjected to irradiation in the head and neck area less than 1 year before implantation.
* Untreated periodontitis.
* Poor oral hygiene and motivation.
* Pregnant or nursing.
* Substance abuse/smoking.
* Psychiatric problems or unrealistic expectations.
* Severe bruxism or clenching.
* Treated or under treatment with intravenous amino-bisphosphonates.
* Lack of opposite occluding dentition/prosthesis in the area intended for implant placement.
* Active infection, current or previous pathology or severe inflammation in the area intended for implant placement.
* Need of bone augmentation procedures at implant placement site.
* Unable to open mouth sufficiently to accommodate the surgical tooling.
* Patients participating in other studies, if the present protocol could not be properly followed.
* Referred only for implant placement or unable to attend a 1-year follow-up.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
bone width and height gain | 4 months
  Bone width and height in millimeter using CBCT

SECONDARY OUTCOMES:
ISQ (Implant Stability Quotients) score secondary implant stability | 6 months
  ISQ using ostell device ( scale from 0-100)